CLINICAL TRIAL: NCT03349281
Title: A Phase I Trial of Pevonedistat in Combination With Induction Chemotherapy for Adolescent and Young Adults With Relapsed/Refractory Acute Lymphoblastic Leukemia or Lymphoblastic Non-Hodgkin Lymphoma
Brief Title: Pevonedistat With VXLD Chemotherapy for Adolescent/Young Adults With Relapsed/Refractory ALL or Lymphoblastic NHL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Julio Barredo, MD (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor-Investigator, Julio Barredo, MD, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170602; X15015 (Other: Takeda)
Record Dates: First submitted 2017-11-07; First posted 2017-11-21 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Refractory Acute Lymphoblastic Leukemia; Relapsed Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pevonedistat; Vincristine; Dexamethasone; Calcium Dobesilate; pegaspargase; Doxorubicin; Cytarabine; Methotrexate; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1: Pevonedistat 15 + VXLD (Experimental): * Pevonedistat: 15 mg/m2 intravenously (IV)
  * Vincristine: 1.5 mg/m2/dose IV push
  * Dexamethasone: 10 mg/m2/day divided twice daily
  * PEG-asparaginase: 2000 IU's/m2/day, capped at maximal dose of 3750 IU's.
  * Doxorubicin: 60 mg/m2/day IV
  * Intrathecal (IT) chemotherapy via injection per protocol:
    * All subjects: Cytarabine 70 mg ;
    * For central nervous system (CNS) negative subjects: Methotrexate 15 mg;
    * For CNS positive subjects (Triple IT Therapy): Cytarabine 30 mg, Methotrexate 15 mg, and Hydrocortisone 15 mg.
  Interventions: Drug: Pevonedistat; Drug: Vincristine; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Hydrocortisone
- Dose Level -1: Pevonedistat 10 + VXLD (Active Comparator): * Pevonedistat: 10 mg/m2 IV
  * Vincristine: 1.5 mg/m2/dose IV push
  * Dexamethasone: 10 mg/m2/day divided twice daily
  * PEG-asparaginase: 2000 IU's/m2/day, capped at maximal dose of 3750 IU's.
  * Doxorubicin: 60 mg/m2/day IV
  * Intrathecal (IT) chemotherapy via injection per protocol:
    * All subjects: Cytarabine 70 mg ;
    * For CNS negative subjects: Methotrexate 15 mg;
    * For CNS positive subjects (Triple IT Therapy): Cytarabine 30 mg, Methotrexate 15 mg, and Hydrocortisone 15 mg.
  Interventions: Drug: Pevonedistat; Drug: Vincristine; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Hydrocortisone
- Dose Level 2: Pevonedistat 20 + VXLD (Active Comparator): * Pevonedistat: 20 mg/m2 IV
  * Vincristine: 1.5 mg/m2/dose IV push
  * Dexamethasone: 10 mg/m2/day divided twice daily
  * PEG-asparaginase: 2000 IU's/m2/day, capped at maximal dose of 3750 IU's.
  * Doxorubicin: 60 mg/m2/day IV
  * Intrathecal (IT) chemotherapy via injection per protocol:
    * All subjects: Cytarabine 70 mg ;
    * For CNS negative subjects: Methotrexate 15 mg;
    * For CNS positive subjects (Triple IT Therapy): Cytarabine 30 mg, Methotrexate 15 mg, and Hydrocortisone 15 mg.
  Interventions: Drug: Pevonedistat; Drug: Vincristine; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Pevonedistat — Administered each cycle on days 1, 3 and 5.
  Other Names: TAK-924; MLN4924
Drug: Vincristine — Administered each cycle on days 2, 9, 16 and 23.
  Other Names: Oncovin; VCR; LCR
Drug: Dexamethasone — Taken orally each cycle on days 2 through 15.
  Other Names: Decadron; Hexadrol; Dexone; Dexameth
Drug: PEG-asparaginase — Administered via intramuscular injection (IM) each cycle on days 9 and 23.
  Other Names: Oncaspar; Pegaspargase; Polyethylene Glycol Conjugated L-asparaginase-H
Drug: Doxorubicin — Administered via IV each cycle on day 2.
  Other Names: Adriamycin
Drug: Cytarabine — Administered to all subjects via IT injection on day 1; and on days 9, 16, and 23 to CNS positive subjects.
  Other Names: ARA-C
Drug: Methotrexate — Administered via IT injection to CNS negative subjects on day 16; and to CNS positive subjects on days 9, 16 and 23.
  Other Names: MTX; Amethopterin
Drug: Hydrocortisone — Administered via IT injection to CNS positive subjects on days 9, 16, and 23.
  Other Names: Cortisol

SUMMARY:
The investigators postulate that Pevonedistat will be effective in patients with relapsed/refractory acute lymphoblastic leukemia (ALL) when combined with a standard backbone ALL chemotherapy regimen.

DETAILED DESCRIPTION:
This is a phase I study of the addition of pevonedistat to induction chemotherapy for AYA patients (16-39 years of age) with relapsed/refractory ALL utilizing a traditional 3+3 design with dose expansion cohort of 6 patients. Starting dose level for pevonedistat is 15 mg/m2. If the number of dose-limiting toxicities (DLTs) is greater than 1 out of 3 patients in the starting dose level, next dose level is 10 mg/m2 (dose level -1). Chemotherapy will consist of pevonedistat in combination with a standard VXLD regimen. The duration of each cycle will be 29 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 16-39 years of age (AYA).
2. Patients must have a diagnosis of a relapsed / refractory ALL (including induction failure) or lymphoblastic non-hodgkin lymphoma.
3. No known contraindications to intended therapies.
4. Prior anthracycline exposure: Patients must have had less than 450 mg/m2 lifetime exposure of anthracycline chemotherapy. For patients whose cumulative dose is between 350-450 mg/m2, Zinecard is strongly recommended.
5. At least 3 months since the last treatment with a "VXLD" induction/re-induction type regimen (i.e., anthracycline, steroid, asparaginase and vincristine).
6. Eastern Cooperative Oncology Group (ECOG) performance status corresponding to 0, 1, or 2 and / or Karnofsky score above 50%.
7. Clinical laboratory values within the following parameters (repeat if more than 3 days before the first dose):

   1. Albumin > 2.7 g/dL
   2. Total bilirubin ≤ 2.5 x upper limit of normal (ULN).
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN,
   4. Creatinine clearance ≥ 50 mL/min;
   5. White blood cell (WBC) count < 50,000/µL before administration of pevonedistat on Cycle 1 Day 1. Note: Hydroxyurea or leukapheresis may be used to control the level of circulating leukemic blast cell counts. (if applicable)
8. Female patients who:

   * Are postmenopausal (see Appendix for definition) for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential:

     * Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception (see Appendix), at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), or
     * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
9. Male patients, even if surgically sterilized (ie, status postvasectomy), who:

   * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)
10. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
11. Patients must have recovered from the acute side effects of all prior anticancer therapy:

    * At least 1 week from prior cytotoxic chemotherapy.
    * At least 4 weeks from craniospinal irradiation
    * At least 4 months since hematopoietic stem cell transplant (HSCT) with no evidence of acute graft vs host disease (GVHD).

Exclusion Criteria:

1. Treatment with any investigational products within 2 weeks before the first dose of any study drug.
2. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures.
3. Active uncontrolled infection or severe infectious disease, defined as positive blood culture within 48 hours of study registration, need for supplemental oxygen or vasopressors within 48 hours of study entry.
4. Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period.
5. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection.
6. Patients with other malignancies that do not meet the exception in # 5 are excluded from participating in the trial.
7. Life-threatening illness unrelated to cancer.
8. Patients with uncontrolled coagulopathy or bleeding disorder, deemed not to be related to underlying disease.
9. Known human immunodeficiency virus (HIV) seropositive.
10. Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection Note: Patients who have isolated positive hepatitis B core antibody (ie, in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
11. Known hepatic cirrhosis or severe pre-existing hepatic impairment
12. Known cardiopulmonary disease defined as:

    * Unstable angina;
    * Congestive heart failure (New York Heart Association (NYHA) Class III or IV; see appendix);
    * Myocardial infarction (MI) within 6 months prior to first dose (patients who had ischemic heart disease such as a (ACS), MI, and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll);
    * Cardiomyopathy;
    * Clinically significant arrhythmia:

      1. History of polymorphic ventricular fibrillation or torsade de pointes,
      2. Permanent atrial fibrillation [a fib], defined as continuous a fib for ≥ 6 months,
      3. Persistent a fib, defined as sustained a fib lasting > 7 days and/or requiring cardioversion in the 4 weeks before screening,
      4. Grade 3 a fib defined as symptomatic and incompletely controlled medically, or controlled with device (e.g. pacemaker), or ablation and
      5. Patients with paroxysmal a fib or < Gr 3 a fib for period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen.
      6. Implantable cardioverter defibrillator;
      7. Moderate to severe aortic and/or mitral stenosis or other valvulopathy (ongoing);
      8. Clinically significant pulmonary hypertension requiring pharmacologic therapy.
13. Uncontrolled high blood pressure (ie, systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg).
14. Prolonged rate corrected QT (QTc) interval ≥ 500 msec, calculated according to institutional guidelines.
15. Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram or radionuclide angiography.
16. Known moderate to severe chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis.
17. Systemic antineoplastic therapy or radiotherapy for other malignant conditions within 14 days before the first dose of any study drug, except for hydroxyurea.
18. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
19. Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).
20. Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).
21. No systemic corticosteroids allowed aside from dexamethasone treatment directed at leukemia. Systemic corticosteroids used for physiological replacement (e.g., adrenal insufficiency) are allowed.
22. Patients who are allergic to PEG-asparaginase or who cannot tolerate any asparaginase because of history of pancreatitis, will go on study without asparaginase. Substitution for Erwinaze is permitted for patients who had an allergic reaction to PEG-asparaginase.
23. Known intolerance to doxorubicin or vincristine.
24. Patients who have started protocol therapy prior to enrollment. Patient may still enroll if IT therapy was given within 72 hours of study enrollment as part of the diagnostic lumbar procedure.

Ages: 16 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Rate of Toxicity in Study Participants Receiving Protocol Therapy | From Cycle 1 Day 1 to up to 30 days post last dose of protocol therapy, about 90 days
  Rate of study participants receiving Pevonedistat/VXLD therapy who experience dose limiting toxicities (DLTs), serious adverse events (SAEs) and and grade 3 or higher adverse events (AEs). Toxicities will be assessed in terms of nature, grade and attribution to protocol therapy using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03.
Determination of the Maximum Tolerated Dose (MTD) in Study Participants Receiving Protocol Therapy | From Cycle 1 Day 1 to up to 30 days post last dose of protocol therapy, about 90 days
  Determination of the maximum tolerated dose (MTD) of Pevonedistat/VXLD therapy for the purpose of obtaining a recommended phase 2 dose (RP2D) regimen

SECONDARY OUTCOMES:
Rate of Clinical Response in Study Participants Receiving Protocol Therapy | Up to two cycles, about 60 days
  Rate of overall response (complete response (CR) + partial response (PR)) in study participants receiving Pevonedistat/VXLD therapy. Responses will be documented according to International Working Group (IWG) Response Criteria. Morphologic complete remission (CR), cytogenetic CR, and molecular CR will be assessed by blood counts and simultaneous examination of the bone marrow for percentage of bone marrow blasts, as well as cytogenetics and molecular studies of bone marrow mononuclear cells.
Pharmacodynamics (PD): Expression Levels of Endoplasmic Reticulum (ER) Stress Response and Unfolded Protein Response (UPR) in Primary ALL Cells to Pevonedistat Therapy | Cycle 1 Days 1 to 4
  Primary acute lymphoblastic leukemia (ALL) cells will be obtained from peripheral blood and/or bone marrow of study participants. Primary cells will be assayed for cell death and cell cycle using standard methodology. Expression levels of endoplasmic reticulum (ER) stress/unfolded protein response (UPR) will be analyzed. A total of 6 samples will be analyzed to establish the PD of pevonedistat, the first three at the time it is given as a single agent (day 1 window) and the following 3 when given in combination with chemotherapy. A sample will be collected from peripheral blood in Cycle 1 on Day 1 pre-dose (immediately before the administration of pevonedistat), 6 and 24 hours post-dose; and on Day 3 pre-dose, 4, 6 and 24 hours post-dose.
Pharmacokinetics (PK): Maximum (Peak) Plasma Concentration (Cmax) of Pevonedistat | Cycle 1 Days 3 to 6
  Cmax is the maximum (or peak) plasma concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose. Serial blood samples for the determination of plasma concentrations of pevonedistat will be collected at pre-specified time points during Cycle 1 to characterize the PK of pevonedistat in combination with VXLD therapy. Plasma for measuring pevonedistat concentrations will be collected pre-dose on day 3, at the end of infusion (EOI), 30 minutes, 1, 2, 4, 6, 24, 48 and 72 hours post pevonedistat dose (10 PK blood draws in total).
Pharmacokinetics (PK): Single-dose time to reach maximum (peak) concentration (Tmax) of Pevonedistat | Cycle 1 Days 3 to 6
  Tmax is the time it takes a drug or other substance to reach the maximum concentration (Cmax). Serial blood samples for the determination of plasma concentrations of pevonedistat will be collected at pre-specified time points during Cycle 1 to characterize the PK of pevonedistat in combination with VXLD therapy. Plasma for measuring pevonedistat concentrations will be collected pre-dose on day 3, at the end of infusion (EOI), 30 minutes, 1, 2, 4, 6, 24, 48 and 72 hours post pevonedistat dose (10 PK blood draws in total).
Pharmacokinetics (PK): Area Under the Curve (AUC) of Plasma Concentration of Pevonedistat | Cycle 1 Days 3 to 6
  The area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC24hr), and AUC extrapolated to infinity (AUCinf) will be assessed. Serial blood samples for the determination of plasma concentrations of pevonedistat will be collected at pre-specified time points during Cycle 1 to characterize the PK of pevonedistat in combination with VXLD therapy. Plasma for measuring pevonedistat concentrations will be collected pre-dose on day 3, at the end of infusion (EOI), 30 minutes, 1, 2, 4, 6, 24, 48 and 72 hours post pevonedistat dose (10 PK blood draws in total).
Pharmacokinetics (PK): Terminal disposition phase half-life (t1/2) of Plasma Concentration of Pevonedistat | Cycle 1 Days 3 to 6
  Terminal disposition phase half-life (t1/2) will be assessed. Half-life (t1/2) is the amount of time it takes for the drug concentration in the plasma to decline by half. Serial blood samples for the determination of plasma concentrations of pevonedistat will be collected at pre-specified time points during Cycle 1 to characterize the PK of pevonedistat in combination with VXLD therapy. Plasma for measuring pevonedistat concentrations will be collected pre-dose on day 3, at the end of infusion (EOI), 30 minutes, 1, 2, 4, 6, 24, 48 and 72 hours post pevonedistat dose (10 PK blood draws in total).

CONTACTS AND LOCATIONS:
Overall Officials: Julio Barredo, MD, Study Chair — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No